CLINICAL TRIAL: NCT02927951
Title: A Randomized, Double-blind, Placebo-Controlled, Cross-over Study on the Effect of Pregabalin on Pain Related to Walking in Patients With Diabetic Peripheral Neuropathy
Brief Title: The Effect of Pregabalin on Pain Related to Walking in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Old Dominion University (Other)
Responsible Party: Principal Investigator, Aaron I. Vinik, MD, PhD, Director of Research & Neuroendocrine Unit, Eastern Virginia Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-11-FB-0209
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Peripheral Neuropathy; Nerve Pain
Keywords: Diabetes Mellitus; Peripheral Neuropathy; Diabetic Pain
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus; Peripheral Nervous System Diseases | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregabalin at 150 mg bid (Experimental): Each subject was randomized to the treatment for 6 weeks, followed by a 2 week washout period, and then completed the other arm of the study.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Each subject was randomized to the treatment for 6 weeks, followed by a 2 week washout period, and then completed the other arm of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — 150mg bid
  Other Names: Lyrica
  Arms: pregabalin at 150 mg bid
Drug: Placebo — 150mg bid
  Arms: Placebo

SUMMARY:
The hypothesis of this study is that pregabalin, 150 mg bid, will reduce general daytime pain in patients diagnosed with diabetic peripheral neuropathy and that it will also reduce the level of pain associated with walking. Consequently, it is hypothesized that the reduction in pain will result in an increase in the amount of walking they do during the day, improvements in their gait, balance, risk of falls and sleep patterns.

DETAILED DESCRIPTION:
Pregabalin (LYRICA®) is a potent and specific ligand at the alpha-2-delta subunit of voltage-gated calcium channels. It is currently approved for adjunctive therapy for neuropathic pain conditions. Patients with diabetic peripheral neuropathy suffer from pain in their feet which interferes with their ability to walk which includes less walking, an altered gait, and altered balance. At night the peripheral neuropathy also interferes with their sleep patterns.The hypothesis of this study is that pregabalin, 150 mg bid, will reduce general daytime pain in patients diagnosed with diabetic peripheral neuropathy and that it will also reduce the level of pain associated with walking. Consequently, it is hypothesized that the reduction in pain will result in an increase in the amount of walking they do during the day, improvements in their gait, balance, risk of falls and sleep patterns.Pain and sleep quality will be assessed with questionnaires but objective measurements will be used to assess gait, balance, daytime activities (including walking) and sleep patterns.

Statistical Power Calculations were based on the fact that this is a randomized, double-blind, placebo-controlled, 2-period crossover study to be conducted at a single site. Comparisons will be drawn at baseline, at the completion of each 6 weeks of treatment/placebo arm. The study has been powered at 0.80 for a two-tail analysis with a sensitivity to detect a 30% delta in pain perception in 40 subjects. From previous studies, the cross-over design suggested has achieved significance with 20 patients per group. Forty-four patients will be recruited in total. Significance will be established at an alpha level of 0.05. Both parametric and non parametric correlations will be carried out between the different variables measured and progressive logistic regression to determine the relative contributions of pain relief on the primary and secondary variables being measured in the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with painful, peripheral neuropathy (ages 40-75 years) and type 2 diabetes (n=40).

Exclusion Criteria:

* Active ocular or systemic disease
* Recent or recurrent history of musculoskeletal injury,
* Presence of neurological conditions or idiopathic neuropathy
* History of or vertigo
* Use of an aid while walking or difficulty with standing upright
* Visible tremor or uncorrected visual deficits.
* Presence of type 1 diabetes mellitus (defined as C-peptide < 1 ng/ml or diabetes onset at < 35 years of age in a non-obese patient).
* Presence of diabetic retinopathy that is more severe than "background" level.
* Presence of diabetic nephropathy
* Presence of clinically significant neuropathy that is clearly of non-diabetic origin, e.g. alcoholic or autoimmune.
* Bilateral amputation of lower extremities or foot ulcers involving the great toes.
* Presence of neuroarthropathy (Charcot deformity) is allowable.
* History of major macrovascular events such as myocardial infarction or stroke within the past 6 months.
* Patients with moderate or severe hepatic insufficiency or abnormalities of liver function.
* Presence of significant pedal edema.
* Other serious medical conditions that in the opinion of the investigator, would compromise the subject's participation in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Decrease in fall risk associated with walking assessed with the Physiological Profile Assesment | Up to 6 months
  The falls risk will also be ascertained using the long-form Physiological Profile Assessment. The Physiological Profile Assessment has been validated in prospective studies of falls in both community and institutional settings, and predicts those at increased risk of falling with 75-79% accuracy. The Physiological Profile Assessment includes tests of vision (edge contrast sensitivity, high/low contrast visual acuity, depth perception), sensation (ankle touch sensitivity, leg proprioception), leg muscle strength (knee flexion, knee extensors, ankle dorsiflexion), postural sway and postural coordination. Scores from each of these physiologic tests are combined to provide an overall fall risk score that ranges from -2 (very low risk) to +4 (very marked risk).

SECONDARY OUTCOMES:
Patient-assessed change in pain intensity assessed with an 11-point scale | Up to 6 months
  Based on an 11-point scale assessed after walking 50 ft in a laboratory setting.
Sleep quality assessed with the Medical Outcomes Study Sleep Scale questionnaire | Up to 6 months
  assessed at home with the Medical Outcomes Study Sleep Scale questionnaire to be completed in the morning.
Patient Global Impression of Change (PGIC) | Up to 6 months
  Patients will record pain and sleep information in diaries. The Patient Global Impression of Change is a 7-point scale on which patients will rate any change in their overall status that they had experienced since beginning study medication from much improved to much worse. The Patient Global Impression of Change is also a 7-point scale on which the clinician rated the change observed in the patient's overall status since the beginning of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron I Vinik, PhD, MD, Principal Investigator — Eastern Virginia Medical School
Locations (2):
- United States (2):
  - Eastern Virgnia Medical School, Strelitz Diabetes Center, Norfolk, Virginia
  - Strelitz Diabetes Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No